CLINICAL TRIAL: NCT02510755
Title: Stress and Emotional Memory : Functional Neuroanatomy of Post-traumatic Stress Disorder in Adolescents
Brief Title: Stress and Emotional Memory
Acronym: SEME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-035
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTSD group (Other): PTSD group
  Interventions: Other: MRI
- Healthy Volunteers (Other): Healthy Volunteers, age-matched controls.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI

SUMMARY:
A broad group of disorders is associated with severe stress existence in children or adolescents. The most characteristic result, and one of the most serious being the state of post-traumatic stress disorder (PTSD), whose main source consists of physical or sexual violence, and to a lesser extent, accidents public road or natural disaster, whose child was the subject or witness. PTSD is associated with a deleterious effect on cognition and including the mnemonic operation. The painful reminder of the traumatic event is one of the most disabling symptoms. However, there are many other memory disorders that experimental studies gradually update. They maintain a close link with emotional regulation that disturbed you know if PTSD. However the majority of studies on emotion and cognition and their relationship with brain activity took adult subject. Work in adolescents are few on the morphological study, on rare neurobehavioral and reduced to two studies of functional neuroimaging. Contrary to what is observed in adults, morphological studies report consistently, no reduction in hippocampal volume. There is no study in the idle state. Two studies in functional MRI, the first highlighted in PTSD patients inhibition of the activity of the anterior cingulate cortex (ACC) to stimuli such as to evoke the trauma, a second reported increased activity in the prefrontal cortex Median (mPFC) in a inhibition. The objective task of our study is to evaluate the impact of psychological trauma on brain structures involved in the emotional component of the memory (amygdala, hippocampus, prefrontal cortex in particular). For this, the investigators will take in 33 adolescents, including patients with posttraumatic symptomatology and matched controls free of trauma age, several neuroimaging exams, anatomical and functional. The functional review will include some rest and another in activation during episodic memory task designed to assess the influence of self-perception on memory impairment observed in patients. The investigators will check, for each group of patients and controls, the involvement of cortical structures in relation to the regulation of emotional memory (CCA, amygdala and hippocampus). The anatomy of the hippocampus benefit specific imaging methods developed in the unit INSERM U923. Endocrine correlates of stress tests will be studied by a fully-traumatic by salivary cortisol sampling.

This research will clarify the mechanisms involved in emotional and memory impairments secondary to psychological trauma, their relationship with self (judgment and self-esteem) and studying their morphological substrates. A longer-term goal is to offer help in the diagnosis and monitoring of young patients with posttraumatic symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 13-18 years
* Informed consent signed by the legal representative and adolescents (e) itself.
* Speaking French as their mother tongue
* patients:subjects with a history of psychological trauma (eg, accidents of public roads (without head trauma), physical or sexual violence) recruited in the care services of hospitals, the diagnosis of chronic PTSD is made using a standardized interview (SCID).
* Healthy controls : subjects who do not have a history of psychological trauma, nor PTSD

Exclusion Criteria:

* ASD, schizophrenia, ADHD
* Head injury with loss of consciousness
* Regular or recent use of alcohol or drugs
* chronic neurological or endocrine disorder
* use of medication that could interfere with the mnemonic or metabolic measurements (psychotropic, hypnotics, anxiolytics, neuroleptics, benzodiazepines, drugs, antiepileptics anti-inflammatory, anti-histamines, central analgesics and muscle relaxants)
* Contraindications to MRI (claustrophobia, metallic object intracorporal)
* Manual Predominance left
* Severe mental retardation evaluated using two subtests from the WISC-IV scales and WAIS III
* Reading Disorders valued using the read speed test

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2012-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Amplitude of the BOLD fMRI signal measured at rest and during cognitive tasks (activation) | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pédopsychiatrie, Caen, France